CLINICAL TRIAL: NCT05650099
Title: Peri-implant Health of Dental Implants in the Posterior Region; an Evaluation After 10 Years
Acronym: Performance
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 11103
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2023-10

CONDITIONS: Missing Teeth
Keywords: Dental implants
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Implants in the posterior region: 126 patients with one or two missing tooth/teeth in the posterior region were treated 10 years ago with dental implant treatment and implant-supported restorations
  Interventions: Device: One or two dental implants (Biomet3I dental implant system) were placed 10 years ago

INTERVENTIONS:
Device: One or two dental implants (Biomet3I dental implant system) were placed 10 years ago — All patients were 10 years ago referred to the Department of Oral and Maxillofacial Surgery (University of Groningen, University Medical Hospital) because of missing posterior teeth and were treated with dental implant placement and implant-supported restorations. Patients will have a regular routine control visit (as part of regular follow-up of these patients)

SUMMARY:
* Background Adaptation of a dental implant and its restoration to the existing anatomy in the region of a missing tooth is presumed to be a reliable procedure. During the follow-up it appears that peri-implant bone level is stable, peri-implant soft tissues are healthy and patients are satisfied with the result. However, the number of 10-years studies on implants in the posterior region of maxilla and mandible is limited and much more studies with longer follow-up periods are needed to confirm the positive outcomes.
* Main research question The primary objective of the study is marginal bone level changes by radiological assessments at 10-years follow-up. Secondary objectives are implant and restoration survival, condition of peri- implant mucosa and patients' satisfaction.
* Design The study design is an observational study of a group of patients which were treated 10 years ago with a dental implant and an implant-supported restoration because of a missing tooth in the posterior region. Outcomes: primary outcome is the change in marginal peri-implant bone level 10 years after placing the definitive restoration. Secondary outcome measures will be implant and restoration survival, peri-implant mucosa health and patients' satisfaction using a questionnaire.
* Expected results Stable peri-implant bone levels, stable peri-implant soft tissue levels, high implant and restoration survival rate and satisfied patients.

DETAILED DESCRIPTION:
The study design is an observational study of a group of 126 patients which were treated 10 years ago with a dental implant and an implant-supported restoration because of a missing tooth in the posterior region.

* Inclusion criteria:
* Patients referred to the department of Oral and Maxillofacial Surgery 10 years ago and treated with a dental implant and an implant-supported restoration because of having a missing tooth in the posterior region. At the time of treatment:
* The patient was 18 years or older;
* The missing tooth was a premolar or molar in maxilla or mandible;
* Sufficient healthy and vital bone to insert a dental implant with a minimum length of 8.5 mm and at least 4.0 mm in diameter with initial stability > 45 Ncm
* The implant site was free from infection;
* Adequate oral hygiene (modified plaque index and modified sulcus bleeding index ≤ 1);
* Sufficient mesio-distal, bucco-lingual, and interocclusal space for placement of an anatomic restoration;
* The patient was capable of understanding and giving informed consent.
* Exclusion criteria at the time of treatment:
* Medical and general contraindications for the surgical procedures;
* Presence of an active and uncontrolled periodontal disease;
* Bruxism;
* Smoking
* A history of local radiotherapy to the head and neck region.

All patients were 10 years ago referred to the Department of Oral and Maxillofacial Surgery (University of Groningen, University Medical Hospital) because of having a missing tooth in the posterior region and were treated with a dental implant. Patients will have a regular routine control visit (as part of regular follow-up of these patients). All data to be collected are part of the routine visit and collected regularly at earlier routine visits, except for the questionnaire. The questionnaire contains a limited number of questions with respect to satisfaction with the function of the implant-supported restoration. If patients are willing to participate (to use their research data and to fill in the questionnaire), they will be asked to give informed consent by signing a form. After signing, they will be included in the 10-years evaluation as participant. The forms will be collected in the CRF and in the medical record it will be noted that patient has signed the informed consent. Data will be collected during the routine control visit; patients will not have an extra visit for data collection.

ELIGIBILITY:
Inclusion Criteria before treatment:

* Patients referred to the department of Oral and Maxillofacial Surgery 10 years ago and treated with a dental implant and an implant-supported restoration because of having a missing tooth in the posterior region. At the time of treatment:
* The patient was 18 years or older;
* The missing tooth was a premolar or molar in maxilla or mandible;
* Sufficient healthy and vital bone to insert a dental implant with a minimum length of 8.5 mm and at least 4.0 mm in diameter with initial stability > 45 Ncm
* The implant site was free from infection;
* Adequate oral hygiene (modified plaque index and modified sulcus bleeding index ≤ 1);
* Sufficient mesio-distal, bucco-lingual, and interocclusal space for placement of an anatomic restoration;
* The patient was capable of understanding and giving informed consent.

Exclusion Criteria at time of treatment:

* Medical and general contraindications for the surgical procedures;
* Presence of an active and uncontrolled periodontal disease;
* Bruxism;
* Smoking
* A history of local radiotherapy to the head and neck region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study design is an observational study of a group of 126 patients which were treated 10 years ago with a dental implant and an implant-supported restoration because of a missing tooth in the posterior region.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Change in peri-implant marginal bone level | Comparison initial radiograph with radiograph after 10 years
  Change in peri-implant marginal bone level along the implant side measured on radiographs in millimetres

SECONDARY OUTCOMES:
Implant survival | 10 years
  Percentage of initially placed of dental implants present after 10 years
Restoration survival | 10 years
  Survival of implant restorations after 10 years
Peri-implant soft tissue health | Status at 10 years
  Health of peri-implant soft tissues after 10 years measured with an ordinal index
Patient satisfaction | Satisfaction at 10 years
  Satisfaction of patients measured with an VAS scale in questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Henny JA Meijer, Prof, Principal Investigator — UMCG Groningen, Netherlands
Locations (1):
- Dept Oral and Maxillofacial Surgery UMCG, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request

REFERENCES:
- [Background] Telleman G, Raghoebar GM, Vissink A, Meijer HJ. Impact of platform switching on inter-proximal bone levels around short implants in the posterior region; 1-year results from a randomized clinical trial. J Clin Periodontol. 2012 Jul;39(7):688-97. doi: 10.1111/j.1600-051X.2012.01887.x. Epub 2012 Apr 29. PMID 22540412
- [Background] Telleman G, Meijer HJ, Vissink A, Raghoebar GM. Short implants with a nanometer-sized CaP surface provided with either a platform-switched or platform-matched abutment connection in the posterior region: a randomized clinical trial. Clin Oral Implants Res. 2013 Dec;24(12):1316-24. doi: 10.1111/clr.12000. Epub 2012 Sep 10. PMID 22957911